CLINICAL TRIAL: NCT05363085
Title: The Effects of Airway Closure, Expiratory Flow Limitation and of a Passive Chest Wall on the Onset of an Uncontrolled Expiration and on Intracranial Pressure. An Observational Clinical Study on Neurosurgical Patients. (The CeRes-CMV Study)
Brief Title: The Cerebral-Respiratory Interaction in Controlled Mechanically Ventilated Neurosurgical Patients. (The CeRes-CMV Study)
Acronym: CeRes-CMV
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Mariangela Pellegrini, Principal Investigator, Uppsala University
Other Study IDs: CeRes-CMV
Record Dates: First submitted 2022-04-27; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Mechanical Ventilation Complication; Neurological Disorder; Lung Injury
MeSH Terms: conditions — Nervous System Diseases; Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood gas analysis sampled daily shortly before respiratory mechanics data recording
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mechanically ventilated neurosurgical patients: Observational study in mechanically ventilated neurosurgical patients
  Interventions: Other: Mechanically ventilated neurosurgical patients

INTERVENTIONS:
Other: Mechanically ventilated neurosurgical patients — Observational study where respiratory variables and intracranial pressure will be measured during mechanical ventilation and during specific respiratory manoeuvres. No intervention is planned.

SUMMARY:
The impact of mechanical ventilation on intracranial perfusion is still not completely clarified. It is often assumed that raising airway pressure will invariably elevate the intracranial pressure, but this is not always the case.

The effects of airway pressure on intracranial pressure can depend on several factors, and among others, an uncontrolled expiration and consequent lung collapse may have an influence on cerebral perfusion.

This study will investigate the incidence and the consequences of an uncontrolled expiration and expiratory lung collapse in critically ill neurosurgical patients during controlled mechanical ventilation.

Electrical impedance tomography measurements , oesophagus and gastric pressure, electrical activity of the diaphragm and intracranial pressure will be acquired in a synchronised manner during controlled mechanical ventilation. Moreover, airway opening pressure, expiratory flow limitation and recruitment/inflation ratio will be determined during controlled mechanical ventilation, on a daily bases until the patient recover his/her own spontaneous breathing.

ELIGIBILITY:
The patients will be included within 48 hours from initiation of mechanical ventilation and insertion of an external ventricular drainage catheter

Inclusion Criteria:

* Age >18 years;
* MV expected for more than 72 hours;
* Not pregnant;
* Informed consent from patient or next of kin.

Exclusion Criteria:

* Previously demonstrated paralysis of the diaphragm or know pathology of the phrenic nerve or neuromuscular disorder,
* Chest tube,
* Patients with clinical conditions that contraindicate the insertion of esophageal/gastric catheters (e.g., esophagus rupture, esophageal bleeding),
* Pacemaker and/or implantable cardioverter defibrillator, these last being a contraindication for EIT.
* Hemicraniectomy. In case of late hemicraniectomy (after patient inclusion), the patient will drop-out from the study.

Relative contraindication: in case of skull base fracture the patient can be included only if oesophageal/gastric and NAVA catheters can be inserted orally.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients recruitment will be kept equally distributed between sexes.
Study Population: Critically ill adult patients affected by acute brain injury (e.g., subarachnoid hemorrhage, subdural hemorrhage, epidural hemorrhage, traumatic brain injury, intracerebral hemorrhage) admitted to the NICU of Uppsala. Consecutive patients will be prospectively screened for eligibility according to inclusion criteria
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
The incidence of lung collapse | during the period of controlled mechanical ventilation, an average of 14 days
  The incidence of an uncontrolled expiration and consequent expiratory lung collapse (determined by expiratory flow limitation, airway opening pressure and expiratory thoracic impedance) increased chest-wall elastance in neurosurgical patients.
Correlation between lung recruitability and intracerebral pressure | during the period of controlled mechanical ventilation, an average of 14 days
  The influence of lung recruitability (determined by recruitment/inflation ratio and changes of thoracic impedance) on intra cerebral pressure in neurosurgical patients.
Correlation between lung collapse and intracerebral pressure | during the period of controlled mechanical ventilation, an average of 14 days
  The correlation between an uncontrolled expiration (determined by expiratory flow limitation, airway opening and expiratory thoracic impedance), increased chest-wall elastance and intracranial pressure in neurosurgical patients.

SECONDARY OUTCOMES:
Intensive care unit (ICU) and hospital length of stay (LOS); | At ICU/hospital discharge, an average of 30 days
  Correlation between lung collapse and LOS
Number of days of mechanical ventilation | At ICU discharge, an average of 20 days
  Correlation between lung collapse and days of mechanical ventilation
90-days mortality from intensive care unit admission | 90 days after hospital discharge
  Correlation between lung collapse and 90-days mortality
30-day and 90-days neurological and functional outcomes | 90 days after hospital discharge
  Correlation between lung collapse and 30-day and 90-days neurological and functional outcomes (Disability Rating Scale, clinical frailty score, Glasgow Outcome Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Mariangela Pellegrini, MD, PhD, Principal Investigator — Uppsala University Hospital, Uppsala University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bencze R, Kawati R, Hanell A, Lewen A, Enblad P, Engquist H, Bjarnadottir KJ, Joensen O, Barrueta Tenhunen A, Freden F, Brochard L, Perchiazzi G, Pellegrini M. Intracranial response to positive end-expiratory pressure is influenced by lung recruitability and gas distribution during mechanical ventilation in acute brain injury patients: a proof-of-concept physiological study. Intensive Care Med Exp. 2025 Apr 14;13(1):43. doi: 10.1186/s40635-025-00750-y. PMID 40229445